CLINICAL TRIAL: NCT04938024
Title: Hmong Microbiome ANd Gout, Obesity, Vitamin C (HMANGO-C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHARM-2020-29354
Record Dates: First submitted 2021-06-14; First posted 2021-06-24 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Hyperuricemia; Gout
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- People with hyperuricemia (HU) or gout without urate-lowering therapy (ULT) (Experimental): Participants with HU or gout who are not treated with ULT will take 500 mg of vitamin C twice daily for 8 weeks.
  Interventions: Dietary Supplement: Vitamin C
- People with hyperuricemia (HU) or gout with urate-lowering therapy (ULT) (Experimental): Participants with HU or gout who are treated with ULT will take 500 mg of vitamin C twice daily for 8 weeks.
  Interventions: Dietary Supplement: Vitamin C
- People without hyperuricemia (HU) or gout without urate-lowering therapy (ULT) (Active Comparator): Participants without HU or gout who are not treated with ULT will take 500 mg of vitamin C twice daily for 8 weeks.
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C is a commercially available over-the-counter food supplement.
  Other Names: L-ascorbic acid

SUMMARY:
Investigators seek to quantify the impact of vitamin C on patient outcomes, including serum urate level, gout-related symptoms, and obesity (measured by BMI) in both healthy Hmong adults and in Hmong patients with hyperuricemia (HU) and/or gout; identify associations between individuals' taxonomic and functional patterns of gut microbiota and its impact on the serum urate-lowering effect of vitamin C; compare taxonomic and functional patterns of gut microbiota between people with HU and/or gout and people without HU and gout; and identify associations between individuals' taxonomic and functional patterns of gut microbiota and self-reported acute gout trigger foods.

DETAILED DESCRIPTION:
Gout, caused by chronic elevation of serum urate (SU), is the most common form of inflammatory arthritis worldwide. About 3.9% of adults in the U.S. suffer from gout and prevalence is even higher in certain ethnicities. Factors that may influence SU include patients' characteristics (gender, weight, renal function, etc.), genetics, and diet. Foods and beverages that have shown positive association with HU and gout are alcohol (particularly beer), purine-rich foods, red meat, seafood, and sugar-sweetened drinks, while inverse association has been found with dairy intake such as skimmed milk and low-calorie yoghurt, coffee and vitamin C. The gut microbiota composition and function have been linked to common chronic human disorders, such as obesity, diabetes, non-alcoholic fatty liver disease, and rheumatoid arthritis. Intestinal microbiota of gout patients were also found highly distinct from healthy individuals in both organismal and functional structures from a small study conducted in China. Strategies to use personal microbiome features to predict glucose response to specific food have been proposed. However, little is known about the impact of microbiota on food and urate-lowering therapy (ULT). The translational significance of a microbiota-guided approach to select appropriate foods and medications that could prevent the elevation of SU for individuals with gout or at high risk for gout is significant. The Hmong are a unique Asian sub-population. Hmong men exhibit a 2-fold higher prevalence of gout, manifesting it earlier in life and experiencing up to 5-fold increased risk of gout-associated complications, compared to non-Hmong in the US. This could lead to higher rates of cardiometabolic diseases (e.g. hypertension, renal disease, type 2 diabetes [T2DM]), which significantly impact morbidity, mortality and healthcare costs. Accordingly, the investigators seek to quantify the impact of vitamin C on patient outcomes, including serum urate level, gout-related symptoms, and obesity (measured by BMI) in both healthy Hmong adults and in Hmong patients with hyperuricemia (HU) and/or gout; identify associations between individuals' taxonomic and functional patterns of gut microbiota and its impact on the serum urate-lowering effect of vitamin C; compare taxonomic and functional patterns of gut microbiota between people with HU and/or gout and people without HU and gout; and identify associations between individuals' taxonomic and functional patterns of gut microbiota and self-reported acute gout trigger foods.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Hmong persons whose both parents are Hmong, with and without hyperuricemia (serum urate (UA) ≥ 6.8 mg/dL ) and/or gout (defined by 2020 American College of Rheumatology Guideline for the Management of Gout) are eligible for the study.
* For those with gout, participants qualify if they have serum UA ≥ 6.8 mg/dL based on the baseline measurement or serum UA < 6.8 mg/dL based on the baseline measurement with at least 1 episode of peripheral joint or bursal swelling, pain, or tenderness (acute gout flare) in their lifetime, (with or without urate-lowering therapy)

Exclusion Criteria:

* Allergy or sensitivity to vitamin C
* Diagnosis/history of:

  * Gastrointestinal surgery including colectomy, ileectomy, and gastrectomy
  * Inflammatory bowel disease
  * Auto-immune disease
  * Type I diabetes mellitus
  * Severe kidney disease (i.e., on dialysis)
  * End-stage liver disease (i.e. cirrhosis)
  * Glucose-6-phosphate dehydrogenase deficiency, (due to increased bleeding risk in those with G6PD deficiency when receiving vitamin C)
* Pregnant or breastfeeding persons
* Current use of:

  * Antibiotics
  * Probiotics supplement
  * Ketogenic diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in serum urate | 8 weeks
  Serum urate levels (mg/dL) will be measured from baseline to end, and the absolute difference will be reported.

SECONDARY OUTCOMES:
Change in Gout Assessment Questionnaire 2.0 score | 8 weeks
  The Gout Assessment Questionnaire 2.0 (GAQ2.0) contains 25 items covering the following domains: gout overall concern, medication side effects, perception of unmet needs, wellbeing during acute gout attack, and concerns during gout attack. Items are rated on a 5-point likert scale. Total scores range from 25 to 125 with higher scores indicating more gout symptoms.
Change in body mass index (BMI) | 8 weeks
  Change in body mass index (BMI) from baseline to end. BMI is calculated as body weight (in kg) divided by height (in cm) squared. BMI is reported in kg/m^2, and the change will be reported as an absolute value.
Change in Swollen Joint Count (44 Joints) | 8 weeks
  Change in gout-related symptoms will be measured from baseline to end using the Swollen Joint Count (44 Joints) post-administration of vitamin C. Scores range from 0-44 with higher scores indicating more swollen joints.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Straka, PharmD, FCCP, Principal Investigator — Univeristy of Minnesota Department of Experimental and Clinical Pharmacology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Wen YF, Culhane-Pera KA, Pergament SL, Moua Y, Vue B, Yang T, Lo M, Sun B, Knights D, Straka RJ. Hmong microbiome ANd Gout, Obesity, Vitamin C (HMANGO-C): A phase II clinical study protocol. PLoS One. 2023 Feb 1;18(2):e0279830. doi: 10.1371/journal.pone.0279830. eCollection 2023. PMID 36724193